CLINICAL TRIAL: NCT00473668
Title: Non-inferiority of One Formulation of GSK Biologicals' DTPw-HBV/Hib to 2 Formulations of GSK Biologicals' DTPw-HBV/Hib With Respect to the Immune Response to the PRP Antigen, When Administered to Healthy Infants at 6, 10, 14 Weeks of Age
Brief Title: Non-inferiority of GSK Biologicals' DTPw-HBV/Hib Compared to Two Formulations of GSK Biologicals' DTPw-HBV/Hib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 104977
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-03

CONDITIONS: Whole Cell Pertussis; Haemophilus Influenzae Type b; Tetanus; Diphtheria; Hepatitis B
Keywords: Hepatitis B; Tetanus; Diphtheria; Pertussis; Haemophilus influenzae type b Vaccines
MeSH Terms: conditions — Haemophilus Infections; Tetanus; Diphtheria; Hepatitis B; Whooping Cough | interventions — Hiberix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (3):
- TRITANRIX-HEPB/HIBERIX KFT. GROUP (Experimental): Subjects, male or female, aged 6 to 8 weeks received 3 doses of Tritanrix™-HepB/Hiberix™ Kft. vaccine, administered intramuscularly in the anterolateral thigh at 6, 10 and 14 weeks of age.
  Interventions: Biological: Zilbrix-Hib
- TRITANRIX-HEPB/HIBERIX LD GROUP (Active Comparator): Subjects, male or female, aged 6 to 8 weeks received 3 doses of Tritanrix™-HepB/Hiberix™ low-dose (LD) formulation vaccine, administered intramuscularly in the anterolateral thigh at 6, 10 and 14 weeks of age.
  Interventions: Biological: Tritanrix™-HepB/ Hiberix™
- TRITANRIX-HEPB/HIBERIX HD GROUP (Active Comparator): Subjects, male or female, aged 6 to 8 weeks received 3 doses of Tritanrix™-HepB/Hiberix™ high-dose (HD) formulation vaccine, administered intramuscularly in the anterolateral thigh at 6, 10 and 14 weeks of age.
  Interventions: Biological: Tritanrix™-HepB/ Hiberix™

INTERVENTIONS:
Biological: Zilbrix-Hib — Intramuscular injection, 1 dose
  Arms: TRITANRIX-HEPB/HIBERIX KFT. GROUP
Biological: Tritanrix™-HepB/ Hiberix™ — Intramuscular injection, 1 dose
  Arms: TRITANRIX-HEPB/HIBERIX HD GROUP; TRITANRIX-HEPB/HIBERIX LD GROUP

SUMMARY:
The purpose of this observer-blind study is to generate immunogenicity data with one formulation of GSK Biologicals' DTPw-HBV/Hib vaccine after the primary vaccination course and to demonstrate non-inferiority of this vaccine as compared to two formulations of GSK Biologicals' DTPw-HBV/Hib vaccine with respect to the anti-PRP antibody response. Additionally to assess the reactogenicity and safety of GSK Biologicals' DTPw-HBV/Hib vaccine. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 and 8 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Administration of one dose of hepatitis B vaccine at birth

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period with the exception of OPV.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the administration of the first vaccine dose, (with the exception of OPV).
* Bacille Calmette-Guérin (BCG) vaccine received after the first 2 weeks of life.
* Hepatitis B vaccine received after the first week of life.
* Previous vaccination against diphtheria, tetanus, pertussis, Haemophilus influenzae or hepatitis B (except hepatitis B at birth).
* History of diphtheria, tetanus, pertussis, Haemophilus influenzae or hepatitis B diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Other conditions which in the opinion of the investigator may potentially interfere with interpretation of study outcomes.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2007-06-01; Primary Completion 2008-01-30 (Actual); Study Completion 2008-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- India (3):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Kolkotta
  - GSK Investigational Site, Varanasi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Chatterjee S, Rego SJ, D'Souza F, Bhatia BD, Collard A, Datta SK, Jacquet JM. The immunogenicity and safety of a reduced PRP-content DTPw-HBV/Hib vaccine when administered according to the accelerated EPI schedule. BMC Infect Dis. 2010 Oct 15;10:298. doi: 10.1186/1471-2334-10-298. PMID 20950457
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104977 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 300 subjects enrolled in the study, one did not receive any vaccination.
Period: Overall Study
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Started | 100 | 100 | 99
Completed | 95 | 89 | 89
Not Completed | 5 | 11 | 10
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Migrated/moved from study area | 3 | 2 | 0
Not completed — Lost to Follow-up | 0 | 4 | 6
Not completed — Other | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group | Total
Number analyzed (Participants) | 100 | 100 | 99 | 299
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 6.3 (0.59) | 6.4 (0.64) | 6.3 (0.51) | 6.3 (0.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 48 | 37 | 124
  Male | 61 | 52 | 62 | 175

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol-phosphate (PRP) Antigens
Description: A seroprotected subject was defined as a subject with anti-PRP concentrations greater than or equal to (≥) 0.15 microgram per milliliter (µg/mL).
Time Frame: At Month 3
Population: The analyses were performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, which included all evaluable for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
Participants | 93 | 84 | 89
Statistical Analysis 1: Comparison: Tritanrix-HepB/Hiberix Kft. Group vs Tritanrix-HepB/Hiberix LD Group; Demonstration of the non-inferiority of Tritanrix™-HepB/Hiberix™ Kft. vaccine compared to Tritanrix™-HepB/Hiberix™ vaccine with respect to the anti-PRP antibody response, after a three-dose primary vaccination course; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if upper limit (UL) of the two-sided 95% confidence interval (CI) for the differences between the two groups in terms of anti-PRP seroprotection (SPR) rates was below (<) 10%; Difference in anti-PRP SPR rate = -1.18, 95% CI 2-sided [-6.39 to 2.84]
Statistical Analysis 2: Comparison: Tritanrix-HepB/Hiberix Kft. Group vs Tritanrix-HepB/Hiberix HD Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in anti-PRP SPR rate = 0, 95% CI 2-sided [-4.16 to 3.99]

2. Secondary Outcome: Number of Seroprotected Subjects Against Hepatitis B Surface Antigen (HBs)
Description: A seroprotected subject is defined as a vaccinated subject with anti-hepatitis B antibody concentration greater than or equal to (≥) 10 milli-international units per milliliter (mIU/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 92 | 85 | 89
Subjects | 92 | 85 | 89

3. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T) Antigen
Description: A seroprotected subject is defined as a vaccinated subject with anti-D and anti-T antibody concentrations greater than or equal to (≥) 0.1 international units per milliliter (IU/mL). Seroprotection was assesed via enzyme-linked immunosorbent assay (ELISA).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
Subjects
  Anti-D | 93 | 85 | 88
  Anti-T | 93 | 85 | 89

4. Secondary Outcome: Number of Seroprotected Subjects Against Diphteria (D) With Antibody Concentrations Above the Cut-off
Description: Seroprotection cut-off values assessed were greater than or equal to (≥) 0.016 international units per milliliter (IU/mL) in the sera of subjects seronegative before vaccination. Concentrations were assessed via neutralization assay on Vero cells.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
Subjects | 93 | 85 | 89

5. Secondary Outcome: Number of Seropositive Subjects Against Polyribosyl-ribitol-phosphate (PRP) Antigens
Description: Seropositivity was defined as antibody concentrations greater than or equal to (≥) 1 microgram/milliliter (µg/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
Subjects | 88 | 80 | 89

6. Secondary Outcome: Number of Seropositive Subjects Against Bordetella Pertussis (BPT) Antigen
Description: A seropositive subject was defined as a vaccinated subject with anti-BPT antibody concentration greater than or equal to (≥) 15 ELISA units (EL.U) per milliliter (EL.U/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
Subjects | 92 | 85 | 88

7. Secondary Outcome: Number of Subjects With Vaccine Response to Bordetella Pertussis (BPT) Antigen
Description: Vaccine response was defined as: for initially seronegative subjects, antibody concentration greater than or equal to (≥) 15 EL.U/mL; and for initially seropositive subjects, antibody concentration ≥ 1 fold the pre-vaccination antibody concentration.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
Subjects | 91 | 84 | 88

8. Secondary Outcome: Concentration of Antibodies Against Polyribosyl-ribitol-phosphate (PRP) Antigens
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in micrograms per milliliter (μg/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
μg/mL | 26.709 [19.161 to 37.232] | 19.583 [14.019 to 27.356] | 40.748 [32.301 to 51.404]

9. Secondary Outcome: Concentration of Antibodies Against Diphtheria (D) and Tetanus (T) Antigens
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
IU/mL
  Anti-D | 2.894 [2.300 to 3.640] | 1.654 [1.357 to 2.016] | 1.756 [1.406 to 2.193]
  Anti-T | 4.740 [3.777 to 5.950] | 2.772 [2.235 to 3.438] | 2.825 [2.316 to 3.447]

10. Secondary Outcome: Concentration of Antibodies Against Hepatitis B Surface Antigen (HBs)
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 92 | 85 | 89
mIU/mL | 781.1 [629.7 to 968.8] | 695.3 [542.1 to 891.7] | 598.2 [477.7 to 749.1]

11. Secondary Outcome: Concentration of Antibodies Against Bordetella Pertussis (BPT) Antigen
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 93 | 85 | 89
EL.U/mL | 63.4 [55.4 to 72.7] | 100.3 [88.4 to 113.7] | 83.7 [73.6 to 95.2]

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-3) follow-up period post-vaccination
Population: The analyses were performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 97 | 96 | 95
Subjects
  Any Pain, Dose 1 | 74 | 69 | 68
  Grade 3 Pain, Dose 1 | 28 | 28 | 17
  Any Redness, Dose 1 | 55 | 58 | 42
  Grade 3 Redness, Dose 1 | 5 | 10 | 4
  Any Swelling, Dose 1 | 63 | 59 | 51
  Grade 3 Swelling, Dose 1 | 16 | 16 | 17
  Any Pain, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Any Pain, Dose 2 | 76 | 64 | 65
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Grade 3 Pain, Dose 2 | 29 | 24 | 14
  Any Redness, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Any Redness, Dose 2 | 54 | 45 | 42
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Grade 3 Redness, Dose 2 | 4 | 6 | 4
  Any Swelling, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Any Swelling, Dose 2 | 60 | 53 | 48
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Grade 3 Swelling, Dose 2 | 20 | 23 | 15
  Any Pain, Dose 3 | 69 | 61 | 53
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 95 | 89 | 89
  Grade 3 Pain, Dose 3 | 23 | 15 | 10
  Any Redness, Dose 3: number analyzed (Participants) | 95 | 89 | 89
  Any Redness, Dose 3 | 53 | 50 | 41
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 95 | 89 | 89
  Grade 3 Redness, Dose 3 | 6 | 5 | 6
  Any Swelling, Dose 3: number analyzed (Participants) | 95 | 89 | 89
  Any Swelling, Dose 3 | 60 | 50 | 40
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 95 | 89 | 89
  Grade 3 Swelling, Dose 3 | 16 | 11 | 11
  Any Pain, Across doses | 87 | 84 | 81
  Grade 3 Pain, Across doses | 46 | 39 | 26
  Any Redness, Across doses | 73 | 74 | 68
  Grade 3 Redness, Across doses | 13 | 16 | 10
  Any Swelling, Across doses | 80 | 76 | 68
  Grade 3 Swelling, Across doses | 32 | 30 | 30

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of any general symptom regardless of intensity grade. Grade 3 Irritability= crying that could not be comforted/prevented normal activity. Grade 3 Drowsiness/Loss of appetite= Drowsiness/Loss of appetite that prevented normal activity. Grade 3 fever = fever above (>) 39.5°C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period post-vaccination
Population: The analyses were performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 96 | 96 | 95
Subjects
  Any Drowsiness, Dose 1 | 42 | 37 | 29
  Grade 3 Drowsiness, Dose 1 | 2 | 3 | 2
  Related Drowsiness, Dose 1 | 35 | 31 | 24
  Any Fever, Dose 1 | 61 | 51 | 33
  Grade 3 Fever, Dose 1 | 0 | 1 | 1
  Related Fever, Dose 1 | 49 | 42 | 26
  Any Irritability, Dose 1 | 62 | 47 | 46
  Grade 3 Irritability, Dose 1 | 8 | 7 | 3
  Related Irritability, Dose 1 | 49 | 38 | 36
  Any Loss of appetite, Dose 1 | 34 | 28 | 20
  Grade 3 Loss of appetite, Dose 1 | 2 | 3 | 1
  Related Loss of appetite, Dose 1 | 31 | 24 | 15
  Any Drowsiness, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Any Drowsiness, Dose 2 | 52 | 41 | 27
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Grade 3 Drowsiness, Dose 2 | 7 | 3 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Related Drowsiness, Dose 2 | 46 | 37 | 26
  Any Fever, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Any Fever, Dose 2 | 45 | 47 | 31
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Grade 3 Fever, Dose 2 | 0 | 1 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Related Fever, Dose 2 | 39 | 40 | 28
  Any Irritability, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Any Irritability, Dose 2 | 57 | 49 | 41
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Grade 3 Irritability, Dose 2 | 9 | 5 | 3
  Related Irritability, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Related Irritability, Dose 2 | 52 | 46 | 38
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Any Loss of appetite, Dose 2 | 36 | 30 | 19
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Grade 3 Loss of appetite, Dose 2 | 3 | 3 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 96 | 93 | 92
  Related Loss of appetite, Dose 2 | 33 | 29 | 18
  Any Drowsiness, Dose 3: number analyzed (Participants) | 95 | 89 | 88
  Any Drowsiness, Dose 3 | 45 | 35 | 24
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Grade 3 Drowsiness, Dose 3 | 6 | 3 | 2
  Related Drowsiness, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Related Drowsiness, Dose 3 | 44 | 35 | 24
  Any Fever, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Any Fever, Dose 3 | 42 | 31 | 29
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Grade 3 Fever, Dose 3 | 0 | 2 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Related Fever, Dose 3 | 41 | 31 | 29
  Any Irritability, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Any Irritability, Dose 3 | 42 | 45 | 33
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Grade 3 Irritability, Dose 3 | 7 | 6 | 4
  Related Irritability, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Related Irritability, Dose 3 | 41 | 45 | 33
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Any Loss of appetite, Dose 3 | 23 | 27 | 25
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Grade 3 Loss of appetite, Dose 3 | 2 | 3 | 1
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 95 | 89 | 95
  Related Loss of appetite, Dose 3 | 23 | 27 | 25
  Any Drowsiness, Across doses | 64 | 58 | 46
  Grade 3 Drowsiness, Across doses | 10 | 8 | 4
  Related Drowsiness, Across doses | 61 | 55 | 42
  Any Fever, Across doses | 77 | 73 | 57
  Grade 3 Fever, Across doses | 0 | 3 | 1
  Related Fever, Across doses | 73 | 68 | 54
  Any Irritability, Across doses | 75 | 69 | 61
  Grade 3 Irritability, Across doses | 17 | 14 | 8
  Related Irritability, Across doses | 72 | 66 | 58
  Any Loss of appetite, Across doses | 55 | 45 | 40
  Grade 3 Loss of appetite, Across doses | 4 | 5 | 2
  Related Loss of appetite, Across doses | 52 | 43 | 36

14. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-30) follow-up period post-vaccination
Population: The analyses were performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 100 | 99 | 100
Subjects | 6 | 4 | 2

15. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (Day 0-Month 3)
Population: The analyses were performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
Number analyzed (Participants) | 100 | 100 | 99
Subjects | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day post-vaccination period (Days 0-3); Unsolicited AEs: during the 31-day post-vaccination period (Days 0-30); SAEs: during the entire study period (Day 0 - Month 3).
Arm/Group | Tritanrix-HepB/Hiberix Kft. Group | Tritanrix-HepB/Hiberix LD Group | Tritanrix-HepB/Hiberix HD Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 87/100 | 84/100 | 81/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tritanrix-HepB/Hiberix Kft. Group (N=100) | Tritanrix-HepB/Hiberix LD Group (N=100) | Tritanrix-HepB/Hiberix HD Group (N=99)
Pain (General disorders) | 87/97 | 84/96 | 81/95
Redness (mm) (General disorders) | 73/97 | 74/96 | 68/95
Swelling (mm) (General disorders) | 80/97 | 76/96 | 68/95
Drowsiness (General disorders) | 64/96 | 58/96 | 46/95
Fever (Axillary) (General disorders) | 77/96 | 73/96 | 57/95
Irritability (General disorders) | 75/96 | 69/96 | 61/95
Loss of appetite (General disorders) | 55/96 | 45/96 | 40/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.